CLINICAL TRIAL: NCT03958994
Title: Improving the Short Term Management of Patients With Dementia Admitted to Hospital
Brief Title: A Systems Approach to Falls and Discharge Planning
Status: Completed | Type: Observational
Sponsor: Bournemouth University (Other)
Responsible Party: Sponsor
Other Study IDs: 1819-IRASMDO
Record Dates: First submitted 2019-05-10; First posted 2019-05-22 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Dementia; Falls; Discharge Planning
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Qualitative interviews — What are the roles of organisational factors, education and policy in shaping the experiences of staff and carers who care for people with dementia?

SUMMARY:
The aim of this study is to generate knowledge on how to improve care for people living with dementia who are in acute hospital. The framework for data collection will be the SHEL [Software (policy) , Hardware (equipment), Environment and Liveware (people)] guidelines. This tool has been chosen for this research because Adams (2008) as well as George, Long, and Vincent (2013) argue that in order to improve care for people with dementia it is important to focus on both wider distal elements like the structural components of an organisation in addition to proximal features like the people factor.

This framework will allow for interview data to be collected on the following:

1. Interactions between patient, carers and staff.
2. Hardware (equipment) used on the ward.
3. Software (paperwork/policy).
4. The hospital environment.

DETAILED DESCRIPTION:
Background: The Care Quality Commission (2016) notes that the Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust (RBCH) has implemented a number of initiatives aimed at improving care given to people with dementia. However, feedback from patients with dementia indicate that improvements are still required (Care Quality Commission, 2016). Therefore, the main aim of this study is to explore how a systems based approach can be used to help with the discharge planning process and the reduction of falls amongst people with dementia by conducting interviews with hospital staff and carers of people with dementia.

Research question: How can a systems perspective contribute to reducing length of stay for people with dementia in an acute hospital through improvements in discharge planning and falls prevention?

Setting: This study will be conducted at the Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust.

Duration:This study is not expected to last longer than three months.

Methods: The researcher will interview hospital staff and carers of people with dementia for a period of approximately thirty minutes. This study will use a hospital systems approach to identify the following: 1) communication and interpersonal strategies used by professionals in the discharge planning process and the reduction of falls, 2) the effectiveness of equipment such as manual handling aides in helping with the discharge planning process and the reduction of falls amongst people with dementia, 3) the impact of policies in the discharge planning process and the reduction of falls, and 4) the influence of the ward environment in helping with the discharge planning process and the reduction of falls. These questions are embedded in Edwards's (1972), Hawkins's (1987) and Zecevic et al.'s (2007) theoretical framework (interactions, environment, policies and equipment).

The findings from this study will be used to inform practice.

ELIGIBILITY:
Inclusion Criteria:

1. Staff (nursing, medical, allied healthcare professionals, support staff) - those who have worked with people who have dementia and are able and willing to provide informed consent.
2. Carers of people with dementia (paid or unpaid) - those who visit the ward regularly and who are able and willing to give informed consent

Exclusion Criteria:

1. Staff (nursing, medical, allied healthcare professionals, support staff)

   * Staff who have not worked with people who have dementia
   * Staff who are unable or unwilling to provide informed consent.
2. Carers of people with dementia

   * People who do not visit patient's on the ward, regularly.
   * People who are unable or unwilling to provide informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hospital staff and carers of people with dementia
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Systems approach interview guide | 3 months
  Hospital staff and carers experiences of caring for patients with dementia.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Nyman, Study Director — Bournemouth University
Locations (1):
- Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust, Bournemouth, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duah-Owusu White M, Vassallo M, Kelly F, Nyman S. Can a systems approach reduce adverse outcomes in patients with dementia in acute settings? (innovative practice). Dementia (London). 2020 May;19(4):1280-1286. doi: 10.1177/1471301217737690. Epub 2017 Nov 3. No abstract available. PMID 29096545
- [Background] Duah-Owusu White, M., Kelly, F., Vassallo, M., & Nyman, S. Using a systems perspective to understand hospital falls among patients with dementia. Aging and Health Research. 2022; 2(4).
- [Background] Duah-Owusu White M, Vassallo M, Kelly F, Nyman S. Two factors that can increase the length of hospital stay of patients with dementia. Rev Esp Geriatr Gerontol. 2022 Nov-Dec;57(6):298-302. doi: 10.1016/j.regg.2022.10.004. Epub 2022 Nov 18. PMID 36411104
- [Background] Duah-Owusu White M, Kelly F. A narrative review of staff views about dementia care in hospital through the lens of a systems framework. J Res Nurs. 2023 Mar;28(2):120-140. doi: 10.1177/17449871221142104. Epub 2022 Dec 29. PMID 37152201
- [Background] Duah-Owusu White M, Kelly F, Vassallo M, Nyman SR. Understanding the hospital discharge planning process for medical patients with dementia. Contemp Nurse. 2023 Aug-Oct;59(4-5):323-333. doi: 10.1080/10376178.2023.2266530. Epub 2023 Nov 30. PMID 37864828